CLINICAL TRIAL: NCT01146483
Title: Drug-drug Interaction Study in Healthy Male Volunteers Following the Administration of Pantoprazole and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CE 09.252
Record Dates: First submitted 2010-05-25; First posted 2010-06-17 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — Rosuvastatin Calcium; Pantoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantoprazole (Active Comparator): two-arm study: 2-period, 2-sequence, cross-over study.Volunteers will be administered either sequence 1 or sequence 2 randomly.
  Interventions: Drug: Rosuvastatin, Pantoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Rosuvastatin, Pantoprazole

INTERVENTIONS:
Drug: Rosuvastatin, Pantoprazole — Rosuvastatin, 10 mg tablets, single dose on the morning
  Concomitant drug: Pantoprazole; 40 mg tablets, 2 single doses administered 1 hour before rosuvastatin and 23 hours after rosuvastatin administration. A placebo is given on the other period as a crossover design study.
  Other Names: Crestor 10 mg; Pantoloc 40 mg

SUMMARY:
This is a single-center, randomized, 2-period, 2-sequence, cross-over study.

DETAILED DESCRIPTION:
Background:

Notions used to describe drug disposition are being reviewed as the roles of drug membrane transporters are being discovered. In the near past, simple biophysical principles - lipophilicity and passive diffusion - were used to explain drug absorption, distribution and elimination. Today, with more than 367 genes known in humans, membrane transporters occupy a much central role.

Rational:

Drug influx/efflux transporters are expressed in various organs with variable activities and their presence increases (influx) or decreases (efflux) the intracellular concentration of a drug in a specific organ. Therefore, intersubject variability in the activity of these transporters due to genetic polymorphisms or concomitant drug treatments can explain intersubject variability in drug actions.

Rosuvastatin is an HMG-CoA reductase inhibitor and a substrate of OATPs and BCRP. There is not much information on the transporter-mediated disposition of rosuvastatin. Literature suggests that rosuvastatin is a transporter substrate of the influx OATP1B1, 1B3 and 2B1 as well as the efflux BCRP. The efflux of rosuvastatin by BCRP would be of major importance in the hepatocytes. BCRP would be responsible of the excretion of 30% of the unchanged drug in the bile. To confirm this hypothesis and identify patients at risk of toxicity with rosuvastatin, we want to perform a drug-drug interactions study with an inhibitor of BCRP namely, pantoprazole. With this approach, we will confirm if rosuvastatin is a real substrate of BCRP as suggested in the literature.

Methodology:

To determine changes induced by the administration of pantoprazole on the pharmacokinetics of rosuvastatin in healthy volunteers 16 healthy volunteers will be administered a single dose of rosuvastatin with and without (placebo) pantoprazole.

Urine and plasma analysis will be performed by LC-MSMS. Pharmacokinetics analysis will be performed. Plasma and urine concentrations of rosuvastatin will be analysed using a noncompartmental method. Pharmacokinetic parameters calculated in this study will be Cmax, Tmax, AUC0-72, AUC0-∞, Kel, T1/2β, CL/F, CLr, and Ae.

ELIGIBILITY:
Inclusion Criteria:

* Vital Signs, EKG and Clinical Laboratory Values within the normal range
* Body mass index (BMI) [20-29kg/m2]
* Caucasian male
* Age between [18-55]
* Healthy by physical exam
* Non or ex-smoker

Exclusion Criteria:

* Presence or history of intolerance or hypersensibility to proton pump inhibitors or HMG-CoA reductase inhibitors.
* Significant illness. History of cardiovascular, kidney, liver or gastrointestinal disease. Presence of cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
* consumption of an investigational product or donation of blood in the previous 28 days preceding the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine changes induced by pantoprazole administration on the pharmacokinetics of rosuvastatin in healthy volunteers. | 2 weeks
  Rosuvastatin will be administered with and without pantoprazole.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Hamet, M.D., Ph.D., Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada